CLINICAL TRIAL: NCT05788328
Title: A PHASE 1, OPEN-LABEL, FIXED-SEQUENCE STUDY TO ESTIMATE THE EFFECT OF PF-07081532 ADMINISTRATION ON THE SINGLE-DOSE PHARMACOKINETICS OF DABIGATRAN AND ROSUVASTATIN IN OVERWEIGHT OR OBESE ADULT PARTICIPANTS
Brief Title: A Drug-Drug Interaction Study to Estimate the Effect of PF-07081532 on the Pharmacokinetics of Dabigatran and Rosuvastatin in Overweight or Obese Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to terminate clinical development of lotiglipron is based on pharmacokinetic data from Phase 1 drug-drug-interaction studies and laboratory measurements of elevated transaminases in these Phase 1 studies as well as a Phase 2 study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3991047
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Dabigatran etexitlate; Rosuvastatin; Molecular Mechanisms of Pharmacological Action; Physiological Effects of Drugs; BCRP substrate; P-gp substrate; Anticoagulant; Antihyperlipidemic
MeSH Terms: interventions — Dabigatran; Rosuvastatin Calcium

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Period 1 (Active Comparator): Participants will receive dabagatrin etexilate (DE) as a single dose
  Interventions: Drug: Dabigatran etexilate (DE)
- Period 2 (Active Comparator): Participants will receive rosuvastatin as a single dose
  Interventions: Drug: Rosuvastatin
- Period 3 (Active Comparator): Participants will receive PF-07081532 daily titrated
  Interventions: Drug: PF-07081532
- Period 4 (Experimental): Participants will receive PF-07081532 daily and DE as a single dose
  Interventions: Drug: Dabigatran etexilate (DE); Drug: PF-07081532
- Period 5 (Experimental): Participants will receive PF-07081532 daily and rosuvastatin as a single dose
  Interventions: Drug: Rosuvastatin; Drug: PF-07081532
- Period 6 (Active Comparator): Participants will receive PF-07081532 daily titrated
  Interventions: Drug: PF-07081532
- Period 7 (Experimental): Participants will receive PF-07081532 daily and DE as a single dose
  Interventions: Drug: Dabigatran etexilate (DE); Drug: PF-07081532
- Period 8 (Experimental): Participants will receive PF-07081532 daily and rosuvastatin as a single dose
  Interventions: Drug: Rosuvastatin; Drug: PF-07081532

INTERVENTIONS:
Drug: Dabigatran etexilate (DE) — Dabigatran etexilate (DE) as oral capsule
  Other Names: Pradaxa
  Arms: Period 1; Period 4; Period 7
Drug: Rosuvastatin — Rosuvastatin as oral tablet
  Other Names: Crestor
  Arms: Period 2; Period 5; Period 8
Drug: PF-07081532 — PF-07081532 as oral tablets
  Other Names: Lotiglipron
  Arms: Period 3; Period 4; Period 5; Period 6; Period 7; Period 8

SUMMARY:
The purpose of the study was to understand the effect of PF-07081532 on the movement of Dabigatran and Rosuvastatin into, though, and out of the body in healthy overweight or obese adult participants. This study also aims to collect data on safety and how tolerable the study medicine is.

The study is seeking for participants who are:

* Male or female who are 18 years of age or older.
* Healthy but are overweight or obese. Participants will receive dabigatran and rosuvastatin as single doses by mouth 3 times during the study. The amount of the study medicine PF-07081532 will be adjusted over time until any interactions are seen.

PF-07081532 is taken daily by mouth in 8 Study Periods while admitted into the study clinic over 53 days. Once discharged from the study clinic, participants will have a follow-up visit 7 to 10 days post last dose of study medicine. Then another follow-up via telephone contact, 28 to 35 days post last dose of study medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy female and male participants must be at least 18 years of age at the time of signing the ICD (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, physical examination, including blood pressure and pulse rate measurement, standard 12-lead ECG and clinical laboratory tests)
2. BMI: ≥25.0 kg/m2 at Screening
3. Stable body weight, defined as <5 kg change (per participant report) for 90 days before Screening

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease
2. Diagnosis of type 1 or type 2 diabetes mellitus or secondary forms of diabetes at Screening
3. History of myocardial infarction, unstable angina, arterial revascularization, mechanical prosthetic heart valve, stroke, New York Association Functional Class II-IV heart failure, or transient ischemic attack within 6 months of Screening
4. Any malignancy not considered cured (except basal cell carcinoma and squamous cell carcinoma of the skin)
5. Personal or family history of MTC or MEN2, or study participants with suspected MTC per the investigator's judgment
6. Acute pancreatitis, a history of repeated episodes of acute pancreatitis, or history of chronic pancreatitis
7. Symptomatic gallbladder disease
8. Medical history or characteristics suggestive of genetic or syndromic obesity or obesity induced by other endocrinological disorders
9. History of depressive disorder or history of other severe psychiatric disorders within the last 2 years from Screening
10. Any lifetime history of a suicide attempt
11. Known medical history of active liver disease, or prior known drug-induced liver injury
12. History of HIV infection
13. Recent history of bleeding, or risks of bleeding, or abnormal coagulation test (INR >1.3) result at Screening
14. Use of prohibited medications
15. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest
16. Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study result
17. Participants with clinical laboratory test abnormalities at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Qps-Mra, Llc, South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 16 participants were enrolled in the study.
Pre-assignment Details: Study had 8 periods and they were conducted sequentially with no washout days between the periods.
Groups:
- All Participants: Participants received Dabigatran etexilate (DE) 150 milligram (mg) as single oral dose on Day 1 of Period 1 followed by Rosuvastatin (ROSU) 10 mg as single dose on Day 1 of Period 2 followed by oral PF-07081532 titrated from 20 mg up to 40 mg once daily (QD) for 8 days in Period 3 followed by DE 150 mg as single oral dose on Day 1 of Period 4 and PF-07081532 80 mg QD orally for 5 days in Period 4. Participants then received ROSU 10 mg as single oral dose on Day 1 of Period 5 and PF-07081532 80 mg QD orally for 4 days in Period 5 followed by oral PF-07081532 titrated from 20 mg up to 240 mg QD for 17 days in Period 6 followed by DE 150 mg as single oral dose on Day 1 of Period 7 and PF-07081532 240 mg QD orally for 2 days in Period 7 followed by ROSU 10 mg as single oral dose on Day 1 of Period 8 and PF-07081532 240 mg QD orally for 4 days in Period 8.There was no washout periods between the study.
Period: Treatment Period 1 (3 Days)
Arm/Group | All Participants
Started | 16
Completed | 16
Not Completed | 0
Period: Treatment Period 2 (4 Days)
Arm/Group | All Participants
Started | 16
Completed | 16
Not Completed | 0
Period: Treatment Period 3 (8 Days)
Arm/Group | All Participants
Started | 16
Completed | 16
Not Completed | 0
Period: Treatment Period 4 (5 Days)
Arm/Group | All Participants
Started | 16
Completed | 15
Not Completed | 1
Not completed — Other | 1
Period: Treatment Period 5 (4 Days)
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0
Period: Treatment Period 6 (17 Days)
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0
Period: Treatment Period 7 (2 Days)
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0
Period: Treatment Period 8 (4 Days)
Arm/Group | All Participants
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- All Participants: Participants received DE 150 mg as single oral dose on Day 1 of Period 1 followed by ROSU 10 mg as single dose on Day 1 of Period 2 followed by oral PF-07081532 titrated from 20 mg up to 40 mg QD for 8 days in Period 3 followed by DE 150 mg as single oral dose on Day 1 of Period 4 and PF-07081532 80 mg QD orally for 5 days in Period 4. Participants then received ROSU 10 mg as single oral dose on Day 1 of Period 5 and PF-07081532 80 mg QD orally for 4 days in Period 5 followed by oral PF-07081532 titrated from 20 mg up to 240 mg QD for 17 days in Period 6 followed by DE 150 mg as single oral dose on Day 1 of Period 7 and PF-07081532 240 mg QD orally for 2 days in Period 7 followed by ROSU 10 mg as single oral dose on Day 1 of Period 8 and PF-07081532 240 mg QD orally for 4 days in Period 8.There was no washout periods between the study.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.00 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time Zero (0) Extrapolated to Infinity (AUCinf) of Total Dabigatran in Period 1, 4 and 7
Description: AUCinf was calculated as AUClast + (Clast/kel), where AUClast is area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast), Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is first-order elimination rate constant.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose of DE on Day 1 of Period 1, 4 and 7
Population: Pharmacokinetic (PK) parameter set included all participants who received at least 1 dose of rosuvastatin, dabigatran etexilate, and/or PF-07081532 and had at least 1 of the PK parameters of interest calculated. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected for Period 1, 4 and 7 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Groups:
- Period 1: DE 150 mg: Participants received DE 150 mg as single oral dose on Day 1 of Period 1.
- Period 4: DE 150 mg + PF-07081532 80 mg QD: Participants received DE 150 mg as single oral dose on Day 1 of Period 4 and PF-07081532 80 mg QD orally from Day 1 to 5 in Period 4.
- Period 7: PF-07081532 240 mg QD + DE 150 mg: Participants received DE 150 mg as single oral dose on Day 1 of Period 7 and PF-07081532 240 mg QD orally from Day 1 to 2 in Period 7.
Arm/Group | Period 1: DE 150 mg | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg
Number analyzed (Participants) | 16 | 15 | 15
nanogram*hour/milliliter (ng*hr/mL) | 1359 (43) | 1195 (38) | 1141 (92)
Statistical Analysis 1: Comparison: Period 1: DE 150 mg vs Period 4: DE 150 mg + PF-07081532 80 mg QD; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 86.50, 90% CI 2-sided [66.05 to 113.29] — Ratio was of test to reference of adjusted geometric means. Reference arm was DE 150mg (Period 1) and test arm was PF-07081532 80mg QD + DE 150mg (Period 4). Ratios (and 90% CIs) were expressed as percentages
Statistical Analysis 2: Comparison: Period 1: DE 150 mg vs Period 7: PF-07081532 240 mg QD + DE 150 mg; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 82.64, 90% CI 2-sided [63.10 to 108.24] — Ratio was of test to reference of adjusted geometric means. Reference arm was DE 150mg (Period 1) and test arm was PF-07081532 240mg QD + DE 150mg (Period 7). Ratios (and 90% CIs) were expressed as percentages

2. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to the Last Measurable Concentration (AUClast) of Total Dabigatran in Period 1, 4 and 7
Description: AUClast was determined using the linear/log trapezoidal method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose of DE on Day 1 of Period 1, 4 and 7
Population: PK parameter set included all participants who received at least 1 dose of rosuvastatin, dabigatran etexilate, and/or PF-07081532 and had at least 1 of the PK parameters of interest calculated. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected for Period 1, 4 and 7 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 1: DE 150 mg | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg
Number analyzed (Participants) | 16 | 15 | 15
ng*hr/mL | 1326 (44) | 1154 (39) | 1089 (97)
Statistical Analysis 1: Comparison: Period 1: DE 150 mg vs Period 4: DE 150 mg + PF-07081532 80 mg QD; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 85.65, 90% CI 2-sided [64.96 to 112.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Period 1: DE 150 mg vs Period 7: PF-07081532 240 mg QD + DE 150 mg; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 80.81, 90% CI 2-sided [61.28 to 106.55] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: AUCinf of Rosuvastatin in Period 2, 5 and 8
Description: as for outcome 1
Time Frame: Pre-dose (0 hour), 1, 2, 3, 4, 5, 6, 8, 10, 14, 24, 48, 72 and 96 hours post dose of ROSU on Day 1 of Period 2, 5 and 8
Population: PK parameter set included all participants who received at least 1 dose of rosuvastatin, dabigatran etexilate, and/or PF-07081532 and had at least 1 of the PK parameters of interest calculated. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected for Period 2, 5 and 8 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Period 2: ROSU 10 mg: Participants received ROSU 10 mg as single dose on Day 1 of Period 2.
- Period 5: ROSU 10mg + PF-07081532 80 mg QD: Participants received ROSU 10 mg as single oral dose on Day 1 of Period 5 and PF-07081532 80 mg QD orally from Day 1 to 4 in Period 5.
- Period 8: PF-07081532 240 mg QD + ROSU 10 mg: Participants received ROSU 10 mg as single oral dose on Day 1 of Period 8 and PF-07081532 240 mg QD orally from Day 1 to 4 in Period 8.
Arm/Group | Period 2: ROSU 10 mg | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 12 | 14 | 13
ng*hr/mL | 26.86 (36) | 67.79 (58) | 63.83 (60)
Statistical Analysis 1: Comparison: Period 2: ROSU 10 mg vs Period 5: ROSU 10mg + PF-07081532 80 mg QD; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 229.11, 90% CI 2-sided [185.23 to 283.37] — Ratio was of test to reference of adjusted geometric means. The reference arm was rosuvastatin 10 mg (Period 2) and test arm was PF-07081532 80 mg QD+rosuvastatin 10 mg (Period 5). The ratios (and 90% CIs) were expressed as percentages
Statistical Analysis 2: Comparison: Period 2: ROSU 10 mg vs Period 8: PF-07081532 240 mg QD + ROSU 10 mg; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 214.73, 90% CI 2-sided [173.38 to 265.94] — Ratio was of test to reference of adjusted geometric means. The reference arm was rosuvastatin 10 mg (Period 2) and test arm was PF-07081532 240 mg QD+rosuvastatin 10 mg (Period 8). The ratios (and 90% CIs) were expressed as percentages

4. Primary Outcome: AUClast of Rosuvastatin in Period 2, 5 and 8
Description: AUClast was determined using the linear/log trapezoidal method.
Time Frame: Pre-dose (0 hour), 1, 2, 3, 4, 5, 6, 8, 10, 14, 24, 48, 72 and 96 hours post dose of ROSU on Day 1 of Period 2, 5 and 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 2: ROSU 10 mg | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 16 | 15 | 15
ng*hr/mL | 29.69 (47) | 63.30 (58) | 69.03 (68)
Statistical Analysis 1: Comparison: Period 2: ROSU 10 mg vs Period 5: ROSU 10mg + PF-07081532 80 mg QD; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 213.05, 90% CI 2-sided [170.46 to 266.29] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Period 2: ROSU 10 mg vs Period 8: PF-07081532 240 mg QD + ROSU 10 mg; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 232.32, 90% CI 2-sided [185.88 to 290.38] — [estimate comment as in outcome 3, analysis 2]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)- All Causalities
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were any untoward medical incidence in a participant during administered study intervention, whether or not these events are related to study intervention. AEs included both serious adverse events (SAEs) and all non-SAEs. An SAE was any untoward medical occurrence at any dose that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity and lastly causes a congenital anomaly/birth defect.
Time Frame: From first dose of study drug up to 28-35 days post last dose of study intervention (maximum up to 76-83 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Period 3: PF-07081532 40 mg QD: Participants received oral PF-07081532 titrated from 20 mg up to 40 mg QD for 8 days in Period 3.
- Period 6: PF-07081532 240 mg QD: Participants received oral PF-07081532 titrated from 20 mg up to 240 mg QD for 17 days in Period 6.
Arm/Group | Period 1: DE 150 mg | Period 2: ROSU 10 mg | Period 3: PF-07081532 40 mg QD | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 6: PF-07081532 240 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 15 | 15 | 15 | 15
Participants | 0 | 0 | 6 | 15 | 6 | 15 | 4 | 9

6. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)
Description: The following laboratory parameters were assessed according to pre-specified criteria for abnormalities: a) hematology; erythrocytes mean corpuscular hemoglobin (picograms per cells ([pg/cells]) (less than[<]0.9*lower limit of normal [LLN]), eosinophils (10^9/Liter [L]), (more than[>]1.2*upper limit of normal [ULN]), prothrombin time (seconds)(>1.1*ULN), prothrombin international normalized ratio(>1.1*ULN); b) clinical chemistry; direct bilirubin(milligram per deciliter [mg/dL])(>1.5*ULN), aspartate aminotransferase(units per litre [U/L]) (>3.0*ULN), alanine aminotransferase(U/L)(> 3.0*ULN), gamma glutamyl transferase(U/L)(> 3.0*ULN), urate (mg/dL)(> 1.2*ULN), high density lipoprotein(HDL) cholesterol (mg/dl)(<0.8*LLN) and lipase(U/L)(> 1.5*ULN). Number of participants with any laboratory abnormalities (without regard to baseline abnormality) meeting pre-specified criteria are reported in this outcome measure.
Time Frame: During treatment of the study (maximum up to 48 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. No laboratory blood sample draws were planned in Period 1 and Period 2, thus no laboratory abnormalities data were collected for these 2 periods. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Period 3: PF-07081532 40 mg QD | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 6: PF-07081532 240 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 16 | 3 | 15 | 15 | 15 | 15
Participants | 2 | 1 | 1 | 2 | 3 | 15

7. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital signs measurement included blood pressure (systolic blood pressure [SBP], diastolic blood pressure [DBP] and pulse rate (PR) and were measured in a supine position after approximately 5 minutes of rest for the participant. Clinical significance in vital signs was judged by investigator.
Time Frame: From first dose of study drug up to 28-35 days post last dose of study intervention (maximum up to 76-83 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: DE 150 mg | Period 2: ROSU 10 mg | Period 3: PF-07081532 40 mg QD | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 6: PF-07081532 240 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 1 | 15 | 15 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percent Change From Baseline in Body Weight
Time Frame: Baseline, Day 1 and 8 of Period 3, Day 1 of Period 5, Day 5 and 12 of Period 6, Day 1 and 5 of Period 8 and follow-up (28-35 days post last dose; up to 76 to 83 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable body weight were analyzed and reported under 'All participants' in this outcome measure. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | All Participants
Number analyzed (Participants) | 16
Percent change
  Day 1 of Period 3 | -0.51 (0.950)
  Day 8 of Period 3 | -1.02 (1.559)
  Day 1 of Period 5: number analyzed (Participants) | 15
  Day 1 of Period 5 | -2.58 (2.146)
  Day 5 of Period 6: number analyzed (Participants) | 15
  Day 5 of Period 6 | -3.32 (2.170)
  Day 12 of Period 6: number analyzed (Participants) | 15
  Day 12 of Period 6 | -4.82 (2.276)
  Day 1 of Period 8: number analyzed (Participants) | 15
  Day 1 of Period 8 | -6.52 (3.272)
  Day 5 of Period 8: number analyzed (Participants) | 15
  Day 5 of Period 8 | -6.90 (2.778)
  Follow-up | -6.01 (3.327)

9. Secondary Outcome: Number of Participants With Pre-defined Criteria of Electrocardiogram (ECG) Parameters
Description: Pre-defined criteria for ECG abnormalities included: PR interval aggregate (millisecond [msec], max. >=300; baseline > 200 and max. increase >= 25 percent (%); baseline > 200 and max. increase >= 25%), QRS interval (msec, max >=140; max. increase >= 50%), QT interval correct by Frederica formula (QTCF) interval aggregate (msec, 450 < max <= 480; 480 < max. <= 500; max. > 500; 30 < max. increase <= 60; max. increase > 60). Number of participants with at least 1 ECG abnormality are reported in this outcome measure.
Time Frame: From first dose of study drug up to 28-35 days post last dose of study intervention (maximum up to 76-83 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected for Period 1, 3, 4, 6 and 8 only.
Measure: Count of Participants; unit: Participants
Groups:
- Period 3: PF-07081532 40 mg QD: Participants received oral PF-07081532 titrated from 20 mg up to 40 mg once daily (QD) for 8 days in Period 3.
- Period 6: PF-07081532 240 mg QD: Participants received oral PF-07081532 titrated from 20 mg up to 240 mg once daily (QD) for 17 days in Period 6.
Arm/Group | Period 1: DE 150 mg | Period 3: PF-07081532 40 mg QD | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 6: PF-07081532 240 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 16 | 16 | 1 | 15 | 15
Participants | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants According to Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. Yes/No responses are mapped to Columbia classification algorithm of suicide assessment (C-CASA) categories: completed suicide, suicide attempt, preparatory acts toward imminent suicidal behavior, suicidal ideation, and self-injurious behavior, or no suicidal intent. n this outcome measure, number of participants with positive response (response of "yes") for each of the five categories are reported.
Time Frame: From first dose of study drug up to 28-35 days post last dose of study intervention (maximum up to 76-83 days)
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable C-SSRS were analyzed and reported under 'All participants' in this outcome measure. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 16
Participants
  Day -1 of Period 1 (Completed suicide) | 0
  Day -1 of Period 1 (Suicide attempt) | 0
  Day -1 of Period 1 (Preparatory acts towards imminent suicidal behavior) | 0
  Day -1 of Period 1 (Suicidal ideation) | 0
  Day -1 of Period 1 (Self-injurious behavior, no suicidal intent) | 0
  Day 8 of Period 3 (Completed suicide) | 0
  Day 8 of Period 3 (Suicide attempt) | 0
  Day 8 of Period 3 (Preparatory acts towards imminent suicidal behavior) | 0
  Day 8 of Period 3 (Suicidal ideation) | 0
  Day 8 of Period 3 (Self-injurious behavior, no suicidal intent) | 0
  Day 5 of Period 6 (Completed suicide): number analyzed (Participants) | 15
  Day 5 of Period 6 (Completed suicide) | 0
  Day 5 of Period 6 (Suicide attempt): number analyzed (Participants) | 15
  Day 5 of Period 6 (Suicide attempt) | 0
  Day 5 of Period 6 (Preparatory acts towards imminent suicidal behavior): number analyzed (Participants) | 15
  Day 5 of Period 6 (Preparatory acts towards imminent suicidal behavior) | 0
  Day 5 of Period 6 (Suicidal ideation): number analyzed (Participants) | 15
  Day 5 of Period 6 (Suicidal ideation) | 0
  Day 5 of Period 6 (Self-injurious behavior, no suicidal intent): number analyzed (Participants) | 15
  Day 5 of Period 6 (Self-injurious behavior, no suicidal intent) | 0
  Day 5 of Period 8 (Completed suicide): number analyzed (Participants) | 15
  Day 5 of Period 8 (Completed suicide) | 0
  Day 5 of Period 8 (Suicide attempt): number analyzed (Participants) | 15
  Day 5 of Period 8 (Suicide attempt) | 0
  Day 5 of Period 8 (Preparatory acts towards imminent suicidal behavior): number analyzed (Participants) | 15
  Day 5 of Period 8 (Preparatory acts towards imminent suicidal behavior) | 0
  Day 5 of Period 8 (Suicidal ideation): number analyzed (Participants) | 15
  Day 5 of Period 8 (Suicidal ideation) | 0
  Day 5 of Period 8 (Self-injurious behavior, no suicidal intent): number analyzed (Participants) | 15
  Day 5 of Period 8 (Self-injurious behavior, no suicidal intent) | 0
  Follow-up (Completed suicide) | 0
  Follow-up (Suicide attempt) | 0
  Follow-up (Preparatory acts towards imminent suicidal behavior) | 0
  Follow-up (Suicidal ideation) | 0
  Follow-up (Self-injurious behavior, no suicidal intent) | 0

11. Secondary Outcome: Number of Participants According to Patient Health Questionnaire-9 (PHQ-9) Classification
Description: The PHQ-9 is a 9 item self-report scale for the assessment of depressive symptoms. The questions included "little interest/pleasure in things", "feeling down depressed or hopeless", "trouble falling or staying asleep", "feeling tired or little energy", "poor appetite or overeating", "feeling bad about yourself", "trouble concentrating on things", "moving slowly or fidgety/restless" and "thoughts you be better off dead". Each item was scored on scale of "not at all" (0), "several days" (1), "more than half the days" (2) to "nearly every day" (3). Total score was obtained by addition of scores for each item and resulted into overall possible score range of 0-27. Higher score = greater severity.
Time Frame: Day 1 prior to treatment (Day -1) in Period 1; Day 8 of Period 3; Days 5 of Period 6; Day 1 and 5 of Period 8; Follow-up: up to 53 to 56 days post last dose of study intervention
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable PHQ-9 were analyzed and reported under 'All participants' in this outcome measure. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants received Dabigatran etexilate (DE ) 150 milligram (mg) as single oral dose on Day 1 of Period 1 followed by Rosuvastatin (ROSU ) 10 mg as single dose on Day 1 of Period 2 followed by oral PF-07081532 titrated from 20 mg up to 40 mg once daily (QD) for 8 days in Period 3 followed by DE 150 mg as single oral dose on Day 1 of Period 4 and PF-07081532 80 mg QD orally for 5 days in Period 4. Participants then received ROSU 10 mg as single oral dose on Day 1 of Period 5 and PF-07081532 80 mg QD orally for 4 days in Period 5 followed by oral PF-07081532 titrated from 20 mg up to 240 mg QD for 17 days in Period 6 followed by DE 150 mg as single oral dose on Day 1 of Period 7 and PF-07081532 240 mg QD orally for 2 days in Period 7 followed by ROSU 10 mg as single oral dose on Day 1 of Period 8 and PF-07081532 240 mg QD orally for 4 days in Period 8.There was no washout periods between the study.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Participants
  Day -1 of Period 1: Little interest/pleasure in things: Not at all | 16
  Day -1 of Period 1: Little interest/pleasure in things: Several days | 0
  Day -1 of Period 1: Little interest/pleasure in things: More than half the days | 0
  Day -1 of Period 1: Little interest/pleasure in things: Nearly every day | 0
  Day -1 of Period 1: Feeling down depressed or hopeless: Not at all | 16
  Day -1 of Period 1: Feeling down depressed or hopeless: Several days | 0
  Day -1 of Period 1: Feeling down depressed or hopeless: More than half the days | 0
  Day -1 of Period 1: Feeling down depressed or hopeless: Nearly every day | 0
  Day -1 of Period 1: Trouble falling or staying asleep: Not at all | 15
  Day -1 of Period 1: Trouble falling or staying asleep: Several days | 1
  Day -1 of Period 1: Trouble falling or staying asleep: More than half the days | 0
  Day -1 of Period 1: Trouble falling or staying asleep: Nearly every day | 0
  Day -1 of Period 1: Feeling tired or little energy: Not at all | 16
  Day -1 of Period 1: Feeling tired or little energy: Several days | 0
  Day -1 of Period 1: Feeling tired or little energy: More than half the days | 0
  Day -1 of Period 1: Feeling tired or little energy: Nearly every day | 0
  Day -1 of Period 1: Poor appetite or overeating: Not at all | 16
  Day -1 of Period 1: Poor appetite or overeating: Several days | 0
  Day -1 of Period 1: Poor appetite or overeating: More than half the days | 0
  Day -1 of Period 1: Poor appetite or overeating: Nearly every day | 0
  Day -1 of Period 1: Feeling bad about yourself: Not at all | 16
  Day -1 of Period 1: Feeling bad about yourself: Several days | 0
  Day -1 of Period 1: Feeling bad about yourself: More than half the days | 0
  Day -1 of Period 1: Feeling bad about yourself: Nearly every day | 0
  Day -1 of Period 1: Trouble concentrating on things: Not at all | 15
  Day -1 of Period 1: Trouble concentrating on things: Several days | 1
  Day -1 of Period 1: Trouble concentrating on things: More than half the days | 0
  Day -1 of Period 1: Trouble concentrating on things: Nearly every day | 0
  Day -1 of Period 1: Moving slowly or fidgety/restless: Not at all | 16
  Day -1 of Period 1: Moving slowly or fidgety/restless: Several days | 0
  Day -1 of Period 1: Moving slowly or fidgety/restless: More than half the days | 0
  Day -1 of Period 1: Moving slowly or fidgety/restless: Nearly every day | 0
  Day -1 of Period 1: Thoughts You be better off dead: Not at all | 16
  Day -1 of Period 1: Thoughts You be better off dead: Several days | 0
  Day -1 of Period 1: Thoughts You be better off dead: More than half the days | 0
  Day -1 of Period 1: Thoughts You be better off dead: Nearly every day | 0
  Day 8 of Period 3: Little interest/pleasure in things: Not at all | 16
  Day 8 of Period 3: Little interest/pleasure in things: Several days | 0
  Day 8 of Period 3: Little interest/pleasure in things: More than half the days | 0
  Day 8 of Period 3: Little interest/pleasure in things: Nearly every day | 0
  Day 8 of Period 3: Feeling down depressed or hopeless: Not at all | 16
  Day 8 of Period 3: Feeling down depressed or hopeless: Several days | 0
  Day 8 of Period 3: Feeling down depressed or hopeless: More than half the days | 0
  Day 8 of Period 3: Feeling down depressed or hopeless: Nearly every day | 0
  Day 8 of Period 3: Trouble falling or staying asleep: Not at all | 15
  Day 8 of Period 3: Trouble falling or staying asleep: Several days | 1
  Day 8 of Period 3: Trouble falling or staying asleep: More than half the days | 0
  Day 8 of Period 3: Trouble falling or staying asleep: Nearly every day | 0
  Day 8 of Period 3: Feeling tired or little energy: Not at all | 16
  Day 8 of Period 3: Feeling tired or little energy: Several days | 0
  Day 8 of Period 3: Feeling tired or little energy: More than half the days | 0
  Day 8 of Period 3: Feeling tired or little energy: Nearly every day | 0
  Day 8 of Period 3: Poor appetite or overeating: Not at all | 15
  Day 8 of Period 3: Poor appetite or overeating: Several days | 1
  Day 8 of Period 3: Poor appetite or overeating: More than half the days | 0
  Day 8 of Period 3: Poor appetite or overeating: Nearly every day | 0
  Day 8 of Period 3: Feeling bad about yourself: Not at all | 16
  Day 8 of Period 3: Feeling bad about yourself: Several days | 0
  Day 8 of Period 3: Feeling bad about yourself: More than half the days | 0
  Day 8 of Period 3: Feeling bad about yourself: Nearly every day | 0
  Day 8 of Period 3: Trouble concentrating on things: Not at all | 15
  Day 8 of Period 3: Trouble concentrating on things: Several days | 1
  Day 8 of Period 3: Trouble concentrating on things: More than half the days | 0
  Day 8 of Period 3: Trouble concentrating on things: Nearly every day | 0
  Day 8 of Period 3: Moving slowly or fidgety/restless: Not at all | 16
  Day 8 of Period 3: Moving slowly or fidgety/restless: Several days | 0
  Day 8 of Period 3: Moving slowly or fidgety/restless: More than half the days | 0
  Day 8 of Period 3: Moving slowly or fidgety/restless: Nearly every day | 0
  Day 8 of Period 3: Thoughts you be better off dead: Not at all | 16
  Day 8 of Period 3: Thoughts you be better off dead: Several days | 0
  Day 8 of Period 3: Thoughts you be better off dead: More than half the days | 0
  Day 8 of Period 3: Thoughts you be better off dead: Nearly every day | 0
  Day 5 of Period 6: Little interest/pleasure in things: number analyzed (Participants) | 15
  Day 5 of Period 6: Little interest/pleasure in things: Not at all | 15
  Day 5 of Period 6: Little interest/pleasure in things: Several days | 0
  Day 5 of Period 6: Little interest/pleasure in things: More than half the days | 0
  Day 5 of Period 6: Little interest/pleasure in things: Nearly every day | 0
  Day 5 of Period 6: Feeling down depressed or hopeless: number analyzed (Participants) | 15
  Day 5 of Period 6: Feeling down depressed or hopeless: Not at all | 15
  Day 5 of Period 6: Feeling down depressed or hopeless: Several days | 0
  Day 5 of Period 6: Feeling down depressed or hopeless: More than half the days | 0
  Day 5 of Period 6: Feeling down depressed or hopeless: Nearly every day | 0
  Day 5 of Period 6: Trouble falling or staying asleep: number analyzed (Participants) | 15
  Day 5 of Period 6: Trouble falling or staying asleep: Not at all | 14
  Day 5 of Period 6: Trouble falling or staying asleep: Several days | 1
  Day 5 of Period 6: Trouble falling or staying asleep: More than half the days | 0
  Day 5 of Period 6: Trouble falling or staying asleep: Nearly every day | 0
  Day 5 of Period 6: Feeling tired or little energy: number analyzed (Participants) | 15
  Day 5 of Period 6: Feeling tired or little energy: Not at all | 14
  Day 5 of Period 6: Feeling tired or little energy: Several days | 1
  Day 5 of Period 6: Feeling tired or little energy: More than half the days | 0
  Day 5 of Period 6: Feeling tired or little energy: Nearly every day | 0
  Day 5 of Period 6: Poor appetite or overeating: number analyzed (Participants) | 15
  Day 5 of Period 6: Poor appetite or overeating: Not at all | 8
  Day 5 of Period 6: Poor appetite or overeating: Several days | 4
  Day 5 of Period 6: Poor appetite or overeating: More than half the days | 1
  Day 5 of Period 6: Poor appetite or overeating: Nearly every day | 2
  Day 5 of Period 6: Feeling bad about yourself: number analyzed (Participants) | 15
  Day 5 of Period 6: Feeling bad about yourself: Not at all | 15
  Day 5 of Period 6: Feeling bad about yourself: Several days | 0
  Day 5 of Period 6: Feeling bad about yourself: More than half the days | 0
  Day 5 of Period 6: Feeling bad about yourself: Nearly every day | 0
  Day 5 of Period 6: Trouble concentrating on things: number analyzed (Participants) | 15
  Day 5 of Period 6: Trouble concentrating on things: Not at all | 15
  Day 5 of Period 6: Trouble concentrating on things: Several days | 0
  Day 5 of Period 6: Trouble concentrating on things: More than half the days | 0
  Day 5 of Period 6: Trouble concentrating on things: Nearly every day | 0
  Day 5 of Period 6: Moving slowly or fidgety/restless: number analyzed (Participants) | 15
  Day 5 of Period 6: Moving slowly or fidgety/restless: Not at all | 15
  Day 5 of Period 6: Moving slowly or fidgety/restless: Several days | 0
  Day 5 of Period 6: Moving slowly or fidgety/restless: More than half the days | 0
  Day 5 of Period 6: Moving slowly or fidgety/restless: Nearly every day | 0
  Day 5 of Period 6: Thoughts you be better off dead: number analyzed (Participants) | 15
  Day 5 of Period 6: Thoughts you be better off dead: Not at all | 15
  Day 5 of Period 6: Thoughts you be better off dead: Several days | 0
  Day 5 of Period 6: Thoughts you be better off dead: More than half the days | 0
  Day 5 of Period 6: Thoughts you be better off dead: Nearly every day | 0
  Day 1 of Period 8: PHQ01- Little interest/pleasure in things: number analyzed (Participants) | 15
  Day 1 of Period 8: PHQ01- Little interest/pleasure in things: Not at all | 14
  Day 1 of Period 8: PHQ01- Little interest/pleasure in things: Several days | 1
  Day 1 of Period 8: PHQ01- Little interest/pleasure in things: More than half the days | 0
  Day 1 of Period 8: PHQ01- Little interest/pleasure in things: Nearly every day | 0
  Day 1 of Period 8: Feeling down depressed or hopeless: number analyzed (Participants) | 15
  Day 1 of Period 8: Feeling down depressed or hopeless: Not at all | 15
  Day 1 of Period 8: Feeling down depressed or hopeless: Several days | 0
  Day 1 of Period 8: Feeling down depressed or hopeless: More than half the days | 0
  Day 1 of Period 8: Feeling down depressed or hopeless: Nearly every day | 0
  Day 1 of Period 8: Trouble falling or staying asleep: number analyzed (Participants) | 15
  Day 1 of Period 8: Trouble falling or staying asleep: Not at all | 13
  Day 1 of Period 8: Trouble falling or staying asleep: Several days | 2
  Day 1 of Period 8: Trouble falling or staying asleep: More than half the days | 0
  Day 1 of Period 8: Trouble falling or staying asleep: Nearly every day | 0
  Day 1 of Period 8: Feeling tired or little energy: number analyzed (Participants) | 15
  Day 1 of Period 8: Feeling tired or little energy: Not at all | 11
  Day 1 of Period 8: Feeling tired or little energy: Several days | 3
  Day 1 of Period 8: Feeling tired or little energy: More than half the days | 0
  Day 1 of Period 8: Feeling tired or little energy: Nearly every day | 1
  Day 1 of Period 8: Poor appetite or overeating: number analyzed (Participants) | 15
  Day 1 of Period 8: Poor appetite or overeating: Not at all | 5
  Day 1 of Period 8: Poor appetite or overeating: Several days | 5
  Day 1 of Period 8: Poor appetite or overeating: More than half the days | 1
  Day 1 of Period 8: Poor appetite or overeating: Nearly every day | 4
  Day 1 of Period 8: Feeling bad about yourself: number analyzed (Participants) | 15
  Day 1 of Period 8: Feeling bad about yourself: Not at all | 15
  Day 1 of Period 8: Feeling bad about yourself: Several days | 0
  Day 1 of Period 8: Feeling bad about yourself: More than half the days | 0
  Day 1 of Period 8: Feeling bad about yourself: Nearly every day | 0
  Day 1 of Period 8: Trouble concentrating on things: number analyzed (Participants) | 15
  Day 1 of Period 8: Trouble concentrating on things: Not at all | 14
  Day 1 of Period 8: Trouble concentrating on things: Several days | 1
  Day 1 of Period 8: Trouble concentrating on things: More than half the days | 0
  Day 1 of Period 8: Trouble concentrating on things: Nearly every day | 0
  Day 1 of Period 8: Moving slowly or fidgety/restless: number analyzed (Participants) | 15
  Day 1 of Period 8: Moving slowly or fidgety/restless: Not at all | 14
  Day 1 of Period 8: Moving slowly or fidgety/restless: Several days | 1
  Day 1 of Period 8: Moving slowly or fidgety/restless: More than half the days | 0
  Day 1 of Period 8: Moving slowly or fidgety/restless: Nearly every day | 0
  Day 1 of Period 8: Thoughts you be better off dead: number analyzed (Participants) | 15
  Day 1 of Period 8: Thoughts you be better off dead: Not at all | 15
  Day 1 of Period 8: Thoughts you be better off dead: Several days | 0
  Day 1 of Period 8: Thoughts you be better off dead: More than half the days | 0
  Day 1 of Period 8: Thoughts you be better off dead: Nearly every day | 0
  Day 5 of Period 8: Little interest/pleasure in things: number analyzed (Participants) | 15
  Day 5 of Period 8: Little interest/pleasure in things: Not at all | 14
  Day 5 of Period 8: Little interest/pleasure in things: Several days | 1
  Day 5 of Period 8: Little interest/pleasure in things: More than half the days | 0
  Day 5 of Period 8: Little interest/pleasure in things: Nearly every day | 0
  Day 5 of Period 8: Feeling down depressed or hopeless: number analyzed (Participants) | 15
  Day 5 of Period 8: Feeling down depressed or hopeless: Not at all | 15
  Day 5 of Period 8: Feeling down depressed or hopeless: Several days | 0
  Day 5 of Period 8: Feeling down depressed or hopeless: More than half the days | 0
  Day 5 of Period 8: Feeling down depressed or hopeless: Nearly every day | 0
  Day 5 of Period 8: Trouble falling or staying asleep: number analyzed (Participants) | 15
  Day 5 of Period 8: Trouble falling or staying asleep: Not at all | 13
  Day 5 of Period 8: Trouble falling or staying asleep: Several days | 2
  Day 5 of Period 8: Trouble falling or staying asleep: More than half the days | 0
  Day 5 of Period 8: Trouble falling or staying asleep: Nearly every day | 0
  Day 5 of Period 8: Feeling tired or little energy: number analyzed (Participants) | 15
  Day 5 of Period 8: Feeling tired or little energy: Not at all | 10
  Day 5 of Period 8: Feeling tired or little energy: Several days | 3
  Day 5 of Period 8: Feeling tired or little energy: More than half the days | 0
  Day 5 of Period 8: Feeling tired or little energy: Nearly every day | 2
  Day 5 of Period 8: Poor appetite or overeating: number analyzed (Participants) | 15
  Day 5 of Period 8: Poor appetite or overeating: Not at all | 6
  Day 5 of Period 8: Poor appetite or overeating: Several days | 6
  Day 5 of Period 8: Poor appetite or overeating: More than half the days | 0
  Day 5 of Period 8: Poor appetite or overeating: Nearly every day | 3
  Day 5 of Period 8: Feeling bad about yourself: number analyzed (Participants) | 15
  Day 5 of Period 8: Feeling bad about yourself: Not at all | 15
  Day 5 of Period 8: Feeling bad about yourself: Several days | 0
  Day 5 of Period 8: Feeling bad about yourself: More than half the days | 0
  Day 5 of Period 8: Feeling bad about yourself: Nearly every day | 0
  Day 5 of Period 8: Trouble concentrating on things: number analyzed (Participants) | 15
  Day 5 of Period 8: Trouble concentrating on things: Not at all | 14
  Day 5 of Period 8: Trouble concentrating on things: Several days | 1
  Day 5 of Period 8: Trouble concentrating on things: More than half the days | 0
  Day 5 of Period 8: Trouble concentrating on things: Nearly every day | 0
  Day 5 of Period 8: Moving slowly or fidgety/restless: number analyzed (Participants) | 15
  Day 5 of Period 8: Moving slowly or fidgety/restless: Not at all | 14
  Day 5 of Period 8: Moving slowly or fidgety/restless: Several days | 1
  Day 5 of Period 8: Moving slowly or fidgety/restless: More than half the days | 0
  Day 5 of Period 8: Moving slowly or fidgety/restless: Nearly every day | 0
  Day 5 of Period 8: Thoughts you be better off dead: number analyzed (Participants) | 15
  Day 5 of Period 8: Thoughts you be better off dead: Not at all | 15
  Day 5 of Period 8: Thoughts you be better off dead: Several days | 0
  Day 5 of Period 8: Thoughts you be better off dead: More than half the days | 0
  Day 5 of Period 8: Thoughts you be better off dead: Nearly every day | 0
  Follow-Up: Little interest/pleasure in things: Not at all | 15
  Follow-Up: Little interest/pleasure in things: Several days | 1
  Follow-Up: Little interest/pleasure in things: More than half the days | 0
  Follow-Up: Little interest/pleasure in things: Nearly every day | 0
  Follow-up: Feeling down depressed or hopeless: Not at all | 16
  Follow-up: Feeling down depressed or hopeless: Several days | 0
  Follow-up: Feeling down depressed or hopeless: More than half the days | 0
  Follow-up: Feeling down depressed or hopeless: Nearly every day | 0
  Follow-up: Trouble falling or staying asleep: Not at all | 15
  Follow-up: Trouble falling or staying asleep: Several days | 1
  Follow-up: Trouble falling or staying asleep: More than half the days | 0
  Follow-up: Trouble falling or staying asleep: Nearly every day | 0
  Follow-up: Feeling tired or little energy: Not at all | 15
  Follow-up: Feeling tired or little energy: Several days | 1
  Follow-up: Feeling tired or little energy: More than half the days | 0
  Follow-up: Feeling tired or little energy: Nearly every day | 0
  Follow-up: Poor appetite or overeating: Not at all | 11
  Follow-up: Poor appetite or overeating: Several days | 3
  Follow-up: Poor appetite or overeating: More than half the days | 1
  Follow-up: Poor appetite or overeating: Nearly every day | 1
  Follow-up: Feeling bad about yourself: Not at all | 16
  Follow-up: Feeling bad about yourself: Several days | 0
  Follow-up: Feeling bad about yourself: More than half the days | 0
  Follow-up: Feeling bad about yourself: Nearly every day | 0
  Follow-up: Trouble concentrating on things: Not at all | 16
  Follow-up: Trouble concentrating on things: Several days | 0
  Follow-up: Trouble concentrating on things: More than half the days | 0
  Follow-up: Trouble concentrating on things: Nearly every day | 0
  Follow-up: Moving slowly or fidgety/restless: Not at all | 16
  Follow-up: Moving slowly or fidgety/restless: Several days | 0
  Follow-up: Moving slowly or fidgety/restless: More than half the days | 0
  Follow-up: Moving slowly or fidgety/restless: Nearly every day | 0
  Follow-up: Thoughts you be better off dead: Not at all | 16
  Follow-up: Thoughts you be better off dead: Several days | 0
  Follow-up: Thoughts you be better off dead: More than half the days | 0
  Follow-up: Thoughts you be better off dead: Nearly every day | 0

12. Secondary Outcome: Maximum Observed Concentration (Cmax) of Total Dabigatran in Period 1, 4 and 7
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose of DE on Day 1 of Period 1, 4 and 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: DE 150 mg | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg
Number analyzed (Participants) | 16 | 15 | 15
ng/mL | 186.0 (54) | 86.01 (48) | 90.18 (104)
Statistical Analysis 1: Comparison: Period 1: DE 150 mg vs Period 4: DE 150 mg + PF-07081532 80 mg QD; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 45.25, 90% CI 2-sided [33.97 to 60.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Period 1: DE 150 mg vs Period 7: PF-07081532 240 mg QD + DE 150 mg; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 47.44, 90% CI 2-sided [35.62 to 63.19] — [estimate comment as in outcome 1, analysis 2]

13. Secondary Outcome: Time for Cmax (Tmax) of Total Dabigatran in Period 1, 4 and 7
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose of DE on Day 1 of Period 1, 4 and 7
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Period 1: DE 150 mg | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg
Number analyzed (Participants) | 16 | 15 | 15
Hours | 3.00 [2.00 to 4.00] | 6.00 [2.00 to 12.0] | 6.00 [3.00 to 8.00]

14. Secondary Outcome: Terminal Half-Life (t1/2) of Total Dabigatran in Period 1, 4 and 7
Description: T1/2 was calculated as loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose of DE on Day 1 of Period 1, 4 and 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Period 1: DE 150 mg | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg
Number analyzed (Participants) | 16 | 15 | 15
Hours | 8.921 (2.8387) | 9.023 (1.3586) | 9.208 (2.0514)

15. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Total Dabigatran in Period 1, 4 and 7
Description: Vz/F was calculated as dose/(AUCinf*kel). AUCinf was calculated as AUClast + (Clast/kel), where AUClast is area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast), Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is first-order elimination rate constant.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose of DE on Day 1 of Period 1, 4 and 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Period 1: DE 150 mg | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg
Number analyzed (Participants) | 16 | 15 | 15
Liters | 1374 (53) | 1618 (48) | 1707 (89)

16. Secondary Outcome: Apparent Oral Clearance (CL/F) of Total Dabigatran in Period 1, 4 and 7
Description: CL/F was calculated as dose/AUCinf. AUCinf was calculated as AUClast + (Clast/kel), where AUClast is area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration (Clast), Clast is the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel is first-order elimination rate constant.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 and 48 hours post dose of DE on Day 1 of Period 1, 4 and 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/Hours
Arm/Group | Period 1: DE 150 mg | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg
Number analyzed (Participants) | 16 | 15 | 15
Liters/Hours | 110.3 (43) | 125.6 (38) | 131.5 (92)

17. Secondary Outcome: Cmax of Rosuvastatin in Period 2, 5 and 8
Time Frame: Pre-dose (0 hour), 1, 2, 3, 4, 5, 6, 8, 10, 14, 24, 48, 72 and 96 hours post dose of ROSU on Day 1 of Period 2, 5 and 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: ROSU 10 mg | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 16 | 15 | 15
ng/mL | 2.230 (63) | 3.951 (70) | 4.964 (88)
Statistical Analysis 1: Comparison: Period 2: ROSU 10 mg vs Period 5: ROSU 10mg + PF-07081532 80 mg QD; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 176.39, 90% CI 2-sided [135.51 to 229.60] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Period 2: ROSU 10 mg vs Period 8: PF-07081532 240 mg QD + ROSU 10 mg; Analysis was performed using mixed effect model with treatment as a fixed effect and participant as a random effect; Test type: Other; Ratio of Adjusted Geometric Means = 221.62, 90% CI 2-sided [170.26 to 288.48] — [estimate comment as in outcome 3, analysis 2]

18. Secondary Outcome: Tmax of Rosuvastatin in Period 2, 5 and 8
Time Frame: Pre-dose (0 hour), 1, 2, 3, 4, 5, 6, 8, 10, 14, 24, 48, 72 and 96 hours post dose of ROSU on Day 1 of Period 2, 5 and 8
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Period 2: ROSU 10 mg | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 16 | 15 | 15
Hours | 5.00 [4.00 to 5.00] | 5.00 [3.00 to 10.0] | 5.00 [3.00 to 6.00]

19. Secondary Outcome: t1/2 of Rosuvastatin in Period 2, 5 and 8
Description: as for outcome 14
Time Frame: Pre-dose (0 hour), 1, 2, 3, 4, 5, 6, 8, 10, 14, 24, 48, 72 and 96 hours post dose of ROSU on Day 1 of Period 2, 5 and 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Period 2: ROSU 10 mg | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 12 | 14 | 13
Hours | 25.40 (9.2472) | 25.52 (16.897) | 19.06 (5.0112)

20. Secondary Outcome: Vz/F of Rosuvastatin in Period 2, 5 and 8
Description: as for outcome 15
Time Frame: Pre-dose (0 hour), 1, 2, 3, 4, 5, 6, 8, 10, 14, 24, 48, 72 and 96 hours post dose of ROSU on Day 1 of Period 2, 5 and 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Period 2: ROSU 10 mg | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 12 | 14 | 13
Liters | 12900 (45) | 4753 (88) | 4171 (63)

21. Secondary Outcome: CL/F of Rosuvastatin in Period 2, 5 and 8
Description: as for outcome 16
Time Frame: Pre-dose (0 hour), 1, 2, 3, 4, 5, 6, 8, 10, 14, 24, 48, 72 and 96 hours post dose of ROSU on Day 1 of Period 2, 5 and 8
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/Hours
Arm/Group | Period 2: ROSU 10 mg | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 12 | 14 | 13
Liters/Hours | 372.5 (36) | 147.4 (58) | 156.5 (60)

22. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Time 24 Hours (AUC24) of PF-07081532 When Co-administered With DE and ROSU in Period 4 and 8 Respectively
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 8, 10, 14 and 24 hours post dose of PF-07081532 in Period 4 and 8
Population: PK parameter set included all participants who received at least 1 dose of rosuvastatin, dabigatran etexilate, and/or PF-07081532 and had at least 1 of the PK parameters of interest calculated. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Data for this outcome measure was planned to be collected for Period 4 and 8 only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 15 | 14
ng*hr/mL | 222000 (59) | 701300 (53)

23. Secondary Outcome: Cmax of PF-07081532 When Co-administered With DE and ROSU in Period 4 and 8 Respectively
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 8, 10, 14 and 24 hours post dose of PF-07081532 in Period 4 and 8
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 15 | 14
ng/mL | 15600 (49) | 42730 (43)

24. Secondary Outcome: Tmax of PF-07081532 When Co-administered With DE and ROSU in Period 4 and 8 Respectively
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 8, 10, 14 and 24 hours post dose of PF-07081532 in Period 4 and 8
Population: as for outcome 22
Measure: Median (Full Range); unit: Hours
Arm/Group | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
Number analyzed (Participants) | 15 | 14
Hours | 6.00 [1.00 to 8.00] | 4.00 [2.00 to 10.0]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28-35 days post last dose of study intervention (maximum up to 76-83 days)
Description: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Arm/Group | Period 1: DE 150 mg | Period 2: ROSU 10 mg | Period 3: PF-07081532 40 mg QD | Period 4: DE 150 mg + PF-07081532 80 mg QD | Period 5: ROSU 10mg + PF-07081532 80 mg QD | Period 6: PF-07081532 240 mg QD | Period 7: PF-07081532 240 mg QD + DE 150 mg | Period 8: PF-07081532 240 mg QD + ROSU 10 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/15 | 0/15 | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 6/16 | 15/16 | 6/15 | 15/15 | 4/15 | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: DE 150 mg (N=16) | Period 2: ROSU 10 mg (N=16) | Period 3: PF-07081532 40 mg QD (N=16) | Period 4: DE 150 mg + PF-07081532 80 mg QD (N=16) | Period 5: ROSU 10mg + PF-07081532 80 mg QD (N=15) | Period 6: PF-07081532 240 mg QD (N=15) | Period 7: PF-07081532 240 mg QD + DE 150 mg (N=15) | Period 8: PF-07081532 240 mg QD + ROSU 10 mg (N=15)
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: DE 150 mg (N=16) | Period 2: ROSU 10 mg (N=16) | Period 3: PF-07081532 40 mg QD (N=16) | Period 4: DE 150 mg + PF-07081532 80 mg QD (N=16) | Period 5: ROSU 10mg + PF-07081532 80 mg QD (N=15) | Period 6: PF-07081532 240 mg QD (N=15) | Period 7: PF-07081532 240 mg QD + DE 150 mg (N=15) | Period 8: PF-07081532 240 mg QD + ROSU 10 mg (N=15)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 2 | 6 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 7 | 0 | 4 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 4 | 7 | 0 | 3 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 6 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 0 | 4 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 2 | 5 | 2 | 3
Early satiety (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT05788328/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/28/NCT05788328/SAP_001.pdf